CLINICAL TRIAL: NCT05773300
Title: Control Population for the Mayo Clinic Adult Congenital Heart Disease Registry
Brief Title: Registry for Mayo Clinic Adult Congenital Heart Disease Control Population
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alexander C. Egbe, Principal Investigator, Mayo Clinic
Other Study IDs: 21-011938; R01HL158517 (NIH)
Record Dates: First submitted 2023-03-10; First posted 2023-03-17 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — 2x1ml Whole Blood, 4x1mL plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This research study is being done to provide comparative data to the Mayo Clinic Adult Congenital Heart Disease Registry.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≤ 30.
* No current cardiac medications.
* Systolic BP ≤ 140 mmHg.
* Diastolic BP ≤ 90 mmHg.
* Capacity to consent.

Exclusion Criteria:

* To be assessed via EMR screening.
* Patient confirmation during screening visit.
* Screening tests as applicable.
* History of cardiovascular disease. eGFR < 30.
* Current orthopedic limitations.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be healthy individuals with no history of cardiovascular disease selected from Mayo Clinic in Rochester, Minnesota.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2022-01-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Peak Oxygen Uptake | 6 Months
  Peak Oxygen Uptake (L/min) : 1.7 ± 0.1
Peak Right Ventricular - Pulmonary Coupling | 6 Months
  Peak Right Ventricular - Pulmonary Coupling: (|%|/mmHg): 0.786 ± 0.065

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Egbe, MBBS, MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No